CLINICAL TRIAL: NCT03806582
Title: Effect of a Higher Blood-pressure on Right Ventricular Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, E.C. Boerma, Dr, Frisius Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TPO 1051
Record Dates: First submitted 2018-10-29; First posted 2019-01-16 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Blood Pressure; Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right | interventions — Norepinephrine

STUDY DESIGN:
Masking Description: open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Active Comparator): intervention with norepinephrine to reach a MAP of 85 mmHg for a maximum duration of 1 hour, observation of the effect on right ventricular function
  Interventions: Drug: Norepinephrine
- control (No Intervention): control group; treatment according to current standards, observation of the effect on right ventricular function

INTERVENTIONS:
Drug: Norepinephrine — intervention with norepinephrine to reach a MAP of 85 mmHg
  Arms: intervention

SUMMARY:
Right ventricular (RV) dysfunction in cardiac surgery is an independent risk factor for morbidity and mortality. Raising the systemic blood pressure with norepinephrine seems to have a positive influence on the right ventricular function in several animal studies. The current study is designed to evaluate the effect of a higher blood pressure on the RV function in post cardiac surgery patients.

DETAILED DESCRIPTION:
Goal: To demonstrate differences in RV function by raising the systemic blood pressure with norepinephrine.

Study design: randomized controlled trial Study population: 78 postoperative cardiac surgery patients admitted at the ICU.

Intervention:

* Group 1: (N=22): RVEF<20% and MAP≤65mmHg. Intervention with norepinephrine to reach a MAP of 85mmHg for a maximum duration of two hours.
* Group 2: (N=22): RVEF <20% and MAP≤65mmHg. Control group: treatment according to current standards. Hypotensive patients are treated with fluids and/or vasopressors to gain a mean arterial pressure (MAP) of 65mmHg.
* Group 3: (N=17): RVEF between ≥20 and <30% and MAP ≤65mmHg. Intervention with norepinephrine to reach a MAP of 85mmHg for a maximum duration of two hours.
* Group 4: (N=17): RVEF between ≥20 and <30% and MAP ≤65mmHg. Control group: treatment according to current standards. Hypotensive patients are treated with fluids and/or vasopressors to gain a mean arterial pressure (MAP) of 65mmHg.

Endpoints: Primary endpoint is the difference between the intervention and the control group in the change over time between baseline and the end of the study period (T4) in RVEF. Secondary endpoints are the echocardiographic parameters of RV and LV contractility, RV end-diastolic pressure, cardiac index, and fluid balance.

ELIGIBILITY:
Inclusion Criteria:

* post operative cardiac surgery patients, full sternotomy
* admission at ICU
* informed consent
* right ventricular monitoring by pulmonary artery catheter.
* RVEF <30% + MAP ≤ 65mmHg

Exclusion Criteria:

* no informed consent
* acute surgery
* Off pump cardiac surgery
* Severe tricuspid insufficiency
* Allergy to norepinephrine
* Severe left ventricular hypertrophy with systolic anterior movement
* Chronic use of alpha-blockers
* Irregulair heart rhythm
* Surgical reasons to maintain a low blood pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
right ventricular ejection fraction | 2 hours postoperative
  Primary endpoint is the difference between the intervention and the control group in the change over time between baseline and the end of the study period (T4) in RVEF.

SECONDARY OUTCOMES:
Echocardiographic | 2 hours postoperative
  Echocardiographic parameters of RV and LV contractility
RV end-diastolic pressure | baseline and 15 minutes postoperatively
  RV end-diastolic pressure pre and post intervention
Cardiac index | 2 hours postoperative
  Difference in cardiac index between intervention and control groups
Fluid balance | 2 hours postoperative
  Difference in fluid balance between intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Boerma, Dr, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No